CLINICAL TRIAL: NCT04952038
Title: Effect of Sleep Disorder on Onset and Progression of Amyotrophic Lateral Sclerosis
Brief Title: Sleep Disorders and the Onset and Progression of ALS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020397
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALS patients with sleep disorder
  Interventions: Behavioral: sleep disorder
- ALS patients without sleep disorder

INTERVENTIONS:
Behavioral: sleep disorder — ALS patients with or without sleep disorder
  Groups: ALS patients with sleep disorder

SUMMARY:
200 cases of ALS patients were collected to explore whether sleep disorders are related to earlier onset age, and whether sleep disorders accelerate the progress of ALS and shorten the survival time of ALS patients.

DETAILED DESCRIPTION:
200 patients with ALS were collected. 1) sleep disorders were assessed by Pittsburgh sleep quality index (PSQI) and Epworth Sleepiness Scale (epworth) at baseline Sleeping Scale，ESS）； 2) Name, age, gender and onset site were collected to explore whether sleep disorders were associated with earlier onset age; 3) The patients' function (ALSFRS-R) at baseline and every 3 months within 2 years were collected, and the end-point time (death and invasive breathing) was recorded to evaluate whether sleep disturbance accelerated the decline of patients' function and shortened their short-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed in the Department of Neurology of the Third Hospital of Beijing Medical University since August 2020. The clinical diagnosis of patients with amyotrophic lateral sclerosis includes: probable and define;
* Informed consent has been signed.

Exclusion Criteria:

* Those who can not cooperate to complete the scale and receive follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed as probable, or definite ALS
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
ALSFERS-R | 2 years
  ALS functional score
end point event | 2 years
  death or invasive breathing

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes